CLINICAL TRIAL: NCT03601442
Title: Managed Access Program (MAP) Cohort Treatment Plan CCTL019B2003I to Provide Access for Patients With Out of Specification Leukapheresis Product and/or Out of Specification Manufactured Tisagenlecleucel (CTL019; Kymriah®)
Brief Title: CTL019 Out of Specification MAP for ALL or DLBCL Patients
Status: Available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CCTL019B2003I
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Acute Lymphoblastic Leukemia (ALL); Diffuse Large B-cell Lymphoma (DLBCL)
Keywords: Acute Lymphoblastic Leukemia; ALL; Pediatric; Diffuse Large b-cell Lymphoma; DLBCL; Adult; Relapse; Refractory; CTL019; tisagenlecleucel; Kymriah; CART19; CART; CAR T cells; Chimeric antigen receptor; Manufacturing; Expanded Access; Out of Specification
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large B-Cell, Diffuse; Recurrence | interventions — tisagenlecleucel

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: CTL019 — CTL019
  Other Names: tisagenlecleucel; Kymriah

SUMMARY:
Managed Access Program (MAP) to provide access to CTL019, for acute lymphoblastic leukemia (ALL) or diffuse large b-cell lymphoma (DLBCL) patients with out of specification leukapheresis product and/or manufactured tisagenlecleucel out of specification for commercial release.

DETAILED DESCRIPTION:
The purpose of this Managed Access Program (MAP) Treatment Plan is to provide access to CTL019, for acute lymphoblastic leukemia (ALL) or diffuse large b-cell lymphoma (DLBCL) patients with out of specification leukapheresis product and/or manufactured tisagenlecleucel out of specification for commercial release where no overwhelming safety concerns has been identified for manufacture and release of the out of specification product.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this Treatment Plan have to meet all of the following criteria:

1. Patients must be treated at a healthcare facility that has been certified /qualified by Novartis to dispense and administer tisagenlecleucel in line with the tisagenlecleucel Risk Evaluation and Mitigation Strategy (REMS) in the United States (US) or the local Risk Management Plan (RMP).

   - Note that tisagenlecleucel treatment should be initiated under the direction of and supervised by a HCP experienced in the treatment of hematological malignancies and trained for administration and management of patients treated with tisagenlecleucel. The healthcare facility must have tocilizumab for use in the event of cytokine release syndrome and emergency equipment per patient prior to infusion on site and ensure timely access to additional doses of tocilizumab; for detailed requirements refer to the approved local label.
2. Patients must be prescribed tisagenlecleucel in line with the locally approved indications (for the precise indication statements see approved local product label). These may include:

   * pediatric and young adult patients up to and (including) 25 years of age with refractory/relapsed (r/r) acute lymphoblastic leukemia (B-ALL)
   * adult patients with r/r diffuse large B-cell lymphoma (DLBCL)
3. Informed consent must be obtained prior to treatment
4. The incoming apheresis material and/or the final manufactured product is out of specification due to failure to meet acceptance or release specifications

Exclusion Criteria:

Patients eligible for this Treatment Plan must not meet any of the following criteria:

1. Contraindications as per the approved local label or the IB.

Ages: 1 Day to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Locations (145):
- United States (142):
  - Banner MDACC, Gilbert, Arizona
  - University of Arizona Cancer Center, Phoenix, Arizona
  - Banner University of Arizona Medical Center, Phoenix, Arizona
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner Uni Medical Center Tucson, Tucson, Arizona
  - City of Hope National Medical Center Hematology&HematCellTransplant, Duarte, California
  - City of Hope, Duarte, California
  - Children's Hospital Los Angeles CRFB002H2301, Los Angeles, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Mattel Childrens Hospital UCLA, Los Angeles, California
  - University of California at Los Angeles UCLA, Los Angeles, California
  - Lucile Packard Children s Hospital Stanford University, Palo Alto, California
  - Lucile Packard Childrens Hospital, Palo Alto, California
  - Stanford University Medical Center, Palo Alto, California
  - UC San Diego, San Diego, California
  - University of California at San Diego, Moores Cancer Ctr UCSD, San Diego, California
  - Rady Children s Hospital Dept of Oncology, San Diego, California
  - Rady Childrens Hospital, San Diego, California
  - Ucsf Benioff Childrens Hospital Pediatric Hematology Oncology, San Francisco, California
  - University of Califronia San Francisco, San Francisco, California
  - University of California, Los Angeles, Santa Monica, California
  - Stanford Healthcare, Stanford, California
  - Children's Hospital Colorado, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - University of Miami Hospital, Miami, Florida
  - JHMI All Children s Hospital, St. Petersburg, Florida
  - Emory University School of Medicine Emory University (12), Atlanta, Georgia
  - Emory University School of Medicine/Winship Cancer Institute Winship Cancer Center, Atlanta, Georgia
  - Emory University School of Medicine/Winship Cancer Institute, Atlanta, Georgia
  - Children's Healthcare of Atlanta Cellular Therapies Lab, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Ann and Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Northwestern, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - University of CHicago Comer Children's Hospital Regulatory, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Healthwatch Plaza Research Associates, Louisville, Kentucky
  - University of Maryland Medical Center UMMC, Baltimore, Maryland
  - University of Maryland Medical Center, Baltimore, Maryland
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins Outpatient Center, Baltimore, Maryland
  - Johns Hopkins University Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Massachusetts General Hospital DF/HCC institutions, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - MGH Cancer Center MGH Cancer Center, Boston, Massachusetts
  - MGH Cancer Center, Boston, Massachusetts
  - Dana Farber Cancer Institute Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan IRB, Ann Arbor, Michigan
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Michigan Health System, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Moffitt Cancer Center, Detroit, Michigan
  - Wayne State University - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital Henry Ford, Detroit, Michigan
  - University of Minnesota Masonic Childrens Hospital, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo CLinic, Rochester, Minnesota
  - WUSTL Jewish Barnes, St Louis, Missouri
  - Hackensack University Medical Center Hackensack UMC, Hackensack, New Jersey
  - Hackensack University Medical Center Onc Dept, Hackensack, New Jersey
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute Rosewell, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering, New York, New York
  - Memorial Sloan Kettering Cancer Center MSKCC, New York, New York
  - Memorial Sloan Kettering Cancer Center Oncology, New York, New York
  - Columbia University Medical Center New York Presbyterian CUMC Research Pharmacy, New York, New York
  - Columbia University Medical Center New York Presbyterian Neuroendocrine Unit, New York, New York
  - Memorial Sloan Kettering Cancer Center MSKCC (9), New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina Chapel Hill Physician Office Building, Chapel Hill, North Carolina
  - University of North Carolina Health System, Chapel Hill, North Carolina
  - Atrium Heath, Charlotte, North Carolina
  - Duke University Medical Center Dept. of DUMC (4), Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children s Hospital Medical Center, Cincinnati, Ohio
  - Cincinnati Childrens Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc Drug Shipment, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center Univ. Hospitals of Cleveland, Cleveland, Ohio
  - Nationwide Childrens Hospital Center, Columbus, Ohio
  - OSU Wexner MC James CH, Columbus, Ohio
  - The Ohio State University Hospitals Clinic The Ohio State University, Columbus, Ohio
  - The Ohio State University Hospitals Clinic, Columbus, Ohio
  - The Ohio State University Regulatory, Columbus, Ohio
  - The Ohio State University Comprehensive Cancer Center Ohio State UMC James Cancer Ct, Columbus, Ohio
  - Hematology Oncology Center, Inc., Elyria, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - OHSU, Portland, Oregon
  - Childrens Hospital of Philadelphia CTRB 3006, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia Children's Hospital Of Phil(2), Philadelphia, Pennsylvania
  - Children s Hospital of Philadelphia Patient Treatment, Philadelphia, Pennsylvania
  - Children s Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - The Childrens Hospital of Philadelphia Children's Hosp Philadelphia, Philadelphia, Pennsylvania
  - The Childrens Hospital of Philadelphia Pediatric Oncology/Stem Cell T, Philadelphia, Pennsylvania
  - The Childrens Hospital of Philadelphia Regulatory, Philadelphia, Pennsylvania
  - University of Pennsylvania Health System CERL080AUS90, Philadelphia, Pennsylvania
  - Pennsylvania Oncology/Hemotology Dept.ofPenn. Onc./Hem., Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Medical University of South Carolina MUSC, Charleston, South Carolina
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Methodist University Hospital Blood and Marrow Transplant, Memphis, Tennessee
  - Texas Cancer Center ( Medical City Dallas Hospital) TX Cancer Center, Dallas, Texas
  - Univof Texas Southwestern Medical Center, Dept of Pediatrics, Dallas, Texas
  - U of TX Southwestern Medical Center - SimmonsCompCancerCtr Satellite, Dallas, Texas
  - UT Southwestern Medical Center Pediatric Hematology/Onc, Dallas, Texas
  - UT Southwestern Medical Center UT SW Medical Ctr of Dallas, Dallas, Texas
  - Cook Children's, Fort Worth, Texas
  - Texas Children's Hospital Baylor College of Medicine, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Cancer Center Methodist Cancer Center (2), Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - MD Anderson Cancer Center/University of Texas MDACC, Houston, Texas
  - MD Anderson Cancer Center/University of Texas StudyCoordinator:CTKI258A2102, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Methodist Hospital / Methodist Cancer Center Houston Methodist Hospital, Houston, Texas
  - Methodist Healthcare System, San Antonio, Texas
  - Methodist Hospital, San Antonio, Texas
  - University of Utah / Huntsman Cancer Institute Huntsman Cancer Cente, Salt Lake City, Utah
  - Primary Childrens Medical Center Oncology, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - University of Virginia Health Systems UVA, Charlottesville, Virginia
  - VCU Health Systems, MCV, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center Dept. of FHCRC, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics Hematopoietic Stem Cell Lab, Madison, Wisconsin
  - University Wisconsin Children's Hospital, Madison, Wisconsin
  - Childrens Hospital of Wisconsin, Milwaukee, Wisconsin
  - Medical College of Wisconsin Med College of WI (29), Milwaukee, Wisconsin
- Novartis Investigative Site, Murdoch, Western Australia, Australia
- Canada (2):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec